CLINICAL TRIAL: NCT00574730
Title: CHOP/Rituximab Followed by Maintenance Pegylated Interferon-Alpha (PEG Intron)With the Treatment of Patients With Anthracycline Naïve Indolent/Follicular Non-Hodgkin's Lymphoma
Brief Title: CHOP/Rituximab Followed by Maintenance PEG Intron in Treatment of Indolent/Follicular Non-Hodgkin's Lymphoma
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Nebraska (Other)
Collaborators: Schering-Plough (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 0013-01-FB
Record Dates: First submitted 2007-12-12; First posted 2007-12-17 (Estimated); Last update posted 2023-09-14 (Actual); Status verified 2023-09

CONDITIONS: Non-Hodgkins Lymphoma
MeSH Terms: conditions — Lymphoma, Non-Hodgkin | interventions — peginterferon alfa-2b

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Arm 1 (Experimental): Participants will receive 6 cycles of combination chemotherapy with the standard CHOP regimen given in conjunction with rituximab. Cycles are repeated at 21-day intervals for six to eight cycles. Participants achieving at least a partial response to chemotherapy will begin PEG Intron at a dose of 2g/kg/week subcutaneously. PEG Intron treatment will be continued for 12 months in the absence of signs of progressive/recurrent disease, or unacceptable toxicity/intolerance of therapy.
  Interventions: Drug: CHOP/Rituximab; Drug: PEG INTRON

INTERVENTIONS:
Drug: CHOP/Rituximab — Six cycles of CHOP/Rituximab therapy at 21-day intervals. CHOP chemo will be administered on day 1 after rituximab.
  Cyclophosphamide750mg/m2 IV, Doxorubicin 50mg/m2 IV, Vincristine 1.4mg/m2 (max 2mg) IV, Prednisone 100mg PO daily x 5 days Rituximab 375mg/m2
Drug: PEG INTRON — Pegylated Interferon-alpha 2mg/kg/week for 52 weeks

SUMMARY:
This study will assess the toxicity/safety of CHOP chemotherapy given concurrently with rituximab, followed by maintenance PEG Intron in patients with anthracycline naïve indolent non-Hodgkin's lymphoma. This study will also evaluate response rates, time to progression, molecular response, and immunologic parameters related to this treatment.will have an ocular exam prior to treatment.

Patients in this study will receive 6 cycles of combination chemotherapy with the standard CHOP regimen given in conjunction with rituximab. Cycles are repeated at 21-day intervals for six to eight cycles. Patients achieving at least a partial response to chemotherapy will begin PEG Intron at a dose of 2g/kg/week subcutaneously. PEG Intron treatment will be continued for 12 months in the absence of signs of progressive/recurrent disease, or unacceptable toxicity/intolerance of therapy. PEG Intron dosing will be adjusted based on the presence of symptoms or other clinical manifestations of toxicity. Patients will undergo bone marrow evaluation for molecular testing at baseline. Those found to be positive will have repeat assessments performed post induction therapy, and after six months of PEG Intron. Patients will also undergo immunologic evaluation at baseline, post induction therapy, and after six months of PEG Intron. At the end of PEG Intron therapy, patients will have disease reevaluation and then annual data collection for long-term toxicity, duration of response and survival.

DETAILED DESCRIPTION:
This study will assess the toxicity/safety of CHOP chemotherapy given concurrently with rituximab, followed by maintenance PEG Intron in patients with anthracycline naïve indolent non-Hodgkin's lymphoma. This study will also evaluate response rates, time to progression, molecular response, and immunologic parameters related to this treatment. Adult patients with indolent, advanced stage, anthracycline naive NHL requiring treatment may be eligible. Patients must have measurable disease, no severe organ dysfunction, and normal ejection fraction in older patients. Patients also must have adequate hematologic, hepatic and renal function, performance status, and life expectancy of at least 18 months. Patients may not have CNS lymphoma, uncontrolled co-morbid conditions, pregnancy, HIV, and active psychiatric conditions. Additionally, patients may not have had prior hypersensitivity to interferon-alpha, other cancer within 5 years, significant heart disease or myocardial infarction within the last 6 months, and history of thrombosis. Additionally, patients will have an ocular exam prior to treatment.

Patients in this study will receive 6 cycles of combination chemotherapy with the standard CHOP regimen given in conjunction with rituximab. Cycles are repeated at 21-day intervals for six to eight cycles. Patients achieving at least a partial response to chemotherapy will begin PEG Intron at a dose of 2g/kg/week subcutaneously. PEG Intron treatment will be continued for 12 months in the absence of signs of progressive/recurrent disease, or unacceptable toxicity/intolerance of therapy. PEG Intron dosing will be adjusted based on the presence of symptoms or other clinical manifestations of toxicity. Patients will undergo bone marrow evaluation for molecular testing at baseline. Those found to be positive will have repeat assessments performed post induction therapy, and after six months of PEG Intron. Patients will also undergo immunologic evaluation at baseline, post induction therapy, and after six months of PEG Intron. At the end of PEG Intron therapy, patients will have disease reevaluation and then annual data collection for long-term toxicity, duration of response and survival.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with a diagnosis of advanced stage indolent non-Hodgkin's lymphoma expressing the CD20 surface antigen (as measured by immunohistochemistry or flow cytometry on peripheral blood, marrow, or tumor tissue). Specific histologic subtypes which are eligible include follicular small cleaved cell (follicular grade 1) and follicular mixed small cleaved and large cell (follicular grade 2) lymphoma, and small lymphocytic lymphoma. Patients with indolent follicular lymphoma (follicular grades 1 and with areas of diffuse histology and patients with diffuse follicle center cell lymphoma are eligible as long as the diffuse areas are not felt to represent areas of transformation to diffuse large B-cell lymphoma.
2. Patients with bulky stage II (at least one tumor mass >/= 5 cm), or stage III or stage IV disease.
3. Patients with an expected life expectancy of at least 18 months.
4. Karnofsky Performance Status >70 (ECOG 0, 1)
5. No prior anthracycline/anthracenedione-based chemotherapy (e.g., CHOP, CNOP)
6. No prior chemotherapy, immunotherapy, radiotherapy, or investigational therapies within three weeks of study entry. Steroid therapy is allowed only if required for maintenance of another chronic disease (e.g., rheumatoid arthritis)
7. Patients with newly diagnosed, relapsed, or refractory disease are eligible as long as they have symptoms or signs which require treatment in the opinion of the treating physician.
8. Patients must have at least one bi-dimensionally measurable lesion.
9. Patients aged > 60 years, or patients with a history of coronary artery disease, congestive heart failure, hypertension, diabetes, or hyperlipidemia must have an estimated ejection fraction > 0.45 (45%) by MUGA or echocardiography, performed within two months of study entry.
10. Females of childbearing potential must have a negative serum pregnancy test prior to enrollment in the study.
11. Patients without evidence of severe organ dysfunction as determined within two weeks of study entry:

    Hemoglobin > 8 g/dl; Absolute neutrophil count > 1000/; platelets > 100,000 Creatinine < 2.0 mg/dl, Bilirubin < 2.0 mg/dl; AST < 3 x upper normal; ALP < 3 x upper normal (if liver function abnormalities are felt to be due to hepatic involvement by lymphoma, bilirubin < 6 mg/dl; AST < 4 x upper normal; ALP < 4 x upper normal will be accepted).
12. All patients will have a complete eye examination performed by an ophthalmologist at baseline.

14. Patients with negative HBSAg are eligible. In the absence of HBSAg negative results, the following will apply:

1. Patients with positive HBSAg must be further evaluated for potential risk of hepatitis B reactivation (see baseline evaluations). If it is felt that the benefits of rituximab-based therapy outweigh the risks of Hepatitis B reactivation, the patient may be enrolled at the discretion of the investigator and will be referred to gastroenterology for evaluation and possible prophylactic therapy (see baseline evaluations)
2. If the patient requires immediate treatment prior to determination of HBSAg results, and the risk of lymphoma outweighs the potential risk of hepatitis B reactivation, the patient may be enrolled at the discretion of the investigator.

Exclusion Criteria:

1. Active CNS lymphoma.
2. Uncontrolled/poorly controlled serious nonmalignant disease (e.g., uncontrolled diabetes mellitus, hypertension, angina, chronic obstructive pulmonary disease).
3. History of hypersensitivity to interferon-alpha.
4. Active uncontrolled infection.
5. History of any other malignancy (except for treated squamous cell or basal cell carcinoma of the skin, or cervical intra-epithelial neoplasia of the cervix) within the past five years.
6. New York Heart Association class III or IV heart disease
7. Myocardial infarction within the past six months.
8. Major surgery within the past month.
9. Diagnosis of deep vein thrombosis or pulmonary embolism within the past three months.
10. Females who are pregnant or lactating.
11. Females of childbearing age who are unwilling to use appropriate methods of contraception.
12. Active psychiatric conditions (e.g., untreated severe depression or psychosis).
13. Patients with known HIV infection.
14. Patients who are on another protocol involving non-FDA approved biologics or drugs.
15. Vulnerable subjects.

Ages: 19 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2001-05-23 (Actual); Primary Completion 2005-08-01 (Actual); Study Completion 2012-06-07 (Actual)

PRIMARY OUTCOMES:
Time to Treatment Failure/Duration of Response/Time to Treatment Failure/Survival | Treatment failure: registration to treatment discontinuation/withdrawal for progression, death, AE, etc. Progression: registration to progression. Duration of response: evaluation with a CR, CCR or PR to progression. Time to death: registration to death.
  Treatment failure: registration to treatment discontinuation/withdrawal for progression, death, AE, etc. Progression: registration to progression. Duration of response: evaluation with a CR, CCR or PR to progression. Time to death: registration to death.

SECONDARY OUTCOMES:
Biologic/Immunologic Evaluation | Baseline, post induction therapy and after six months of PEG-Intron.
  Patients with follicular NHL will undergo bone marrow evaluation for the presence of the bcl-2 gene rearrangement at baseline. Those found to be positive will have repeat assessments performed post induction therapy and after six months of PEG Intron.

CONTACTS AND LOCATIONS:
Overall Officials: Robert G Bociek, MD, Principal Investigator — University of Nebraska
Locations (1):
- Unversity of Nebraska Medical Center, Omaha, Nebraska, United States